CLINICAL TRIAL: NCT06798350
Title: Clinical Study on the Role of Inflammatory Markers in Patients With Erectile Dysfunction
Status: Not yet recruiting | Type: Observational
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: XJLL-KY-20252014
Record Dates: First submitted 2025-01-23; First posted 2025-01-29 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Erectile Dysfunction, CTCAE
MeSH Terms: conditions — Erectile Dysfunction

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
* Project Title**: Clinical Study on the Role of Inflammatory Markers in Patients with Erectile Dysfunction
* Research Objective**:

To explore the changes in the levels of inflammatory markers in patients with erectile dysfunction (ED), providing scientific evidence for the diagnosis and treatment of ED.

**Study Design**: Retrospective controlled study

* Total Sample Size**:

  150 cases
* Case Selection**:
* Inclusion Criteria for Case Group**:

  1. Males with regular sexual activity;
  2. Age between 18 and 55 years;
  3. Complete medical records;
  4. Completion of the International Index of Erectile Function-5 (IIEF-5), with IIEF-5 score < 22. Cases with an IIEF-5 score < 22 are diagnosed with ED, while the rest are diagnosed as non-ED.
* Inclusion Criteria for Control Group**:

  1. Males with regular sexual activity;
  2. Age between 18 and 55 years; matched with the case group by age difference < 3 years. If multiple volunteers meet the criteria, the one closest in age to the case group is selected;
  3. Complete medical records;
  4. Completion of the International Index of Erectile Function-5 (IIEF-5), with IIEF-5 score ≥ 22.
* Exclusion Criteria**:

  1. Patients with spinal cord injury, neurological diseases, severe heart disease, or a history of penile fibrosis;
  2. Patients undergoing treatment with phosphodiesterase type 5 inhibitors (PDE-5i);
  3. Patients diagnosed with hormonal abnormalities, hyperthyroidism, hypothyroidism, Peyronie's disease, prostatitis, urethritis, or urinary tract infections;
  4. Patients with poor rapid eye movement (REM) sleep quality.
* Efficacy Assessment**:
* Observational Indicators**:

Peripheral blood count, including monocyte count, neutrophil count, lymphocyte count, and biochemical markers such as C-reactive protein.

**Safety Evaluation Indicators**: Reproductive system damage.

**Statistical Methods**: Data analysis will be performed using R software (version 4.1.6). All statistical tests will be two-sided, with P values < 0.05 considered significant. Normality of data will be assessed using the Shapiro-Wilk test. Data with normal distribution will be presented as mean ± standard deviation, and data with non-normal distribution will be presented as median [interquartile range]. Baseline characteristics will be compared using independent sample t-tests, Mann-Whitney U tests, or chi-square/Fisher's exact tests. Multivariate analysis will be conducted using logistic regression to estimate odds ratios (OR) and 95% confidence intervals (CI). Missing data will be handled using appropriate methods based on the data missing mechanism. To control Type I errors, Bonferroni correction will be applied during multiple comparisons. All analysis procedures and code will be documented in detail to ensure the reproducibility of the analysis.

ELIGIBILITY:
Inclusion Criteria:

- Males with regular sexual activity; Age between 18 and 55 years; matched with the case group by age difference < 3 years. If multiple volunteers meet the criteria, the one closest in age to the case group is selected; Complete medical records; Completion of the International Index of Erectile Function-5 (IIEF-5), with IIEF-5 score ≥ 22.

Exclusion Criteria:

- Patients with spinal cord injury, neurological diseases, severe heart disease, or a history of penile fibrosis; Patients undergoing treatment with phosphodiesterase type 5 inhibitors (PDE-5i); Patients diagnosed with hormonal abnormalities, hyperthyroidism, hypothyroidism, Peyronie's disease, prostatitis, urethritis, or urinary tract infections; Patients with poor rapid eye movement (REM) sleep quality.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Inclusion Criteria for Case Group:
  Males with regular sexual activity; Age between 18 and 55 years; Complete medical records; Completion of the International Index of Erectile Function-5 (IIEF-5), with IIEF-5 score < 22. Cases with an IIEF-5 score < 22 are diagnosed with ED, while the rest are diagnosed as non-ED.
  Inclusion Criteria for Control Group:
  Males with regular sexual activity; Age between 18 and 55 years; matched with the case group by age difference < 3 years. If multiple volunteers meet the criteria, the one closest in age to the case group is selected; Complete medical records; Completion of the International Index of Erectile Function-5 (IIEF-5), with IIEF-5 score ≥ 22.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-03-10 (Estimated); Primary Completion 2025-04-10 (Estimated); Study Completion 2025-05-10 (Estimated)

PRIMARY OUTCOMES:
The diagnosis of ED | A retrospective study observing patients approximately 1 month before and after diagnosis.
  The diagnosis of ED is based on the IIEF-5 questionnaire score, with patients scoring <22 being diagnosed with ED, and the remaining patients being diagnosed as non-ED.